CLINICAL TRIAL: NCT03749863
Title: Safety and Efficacy of Serial Platelet-Rich Plasma Injections for Treatment of Vocal Fold Atrophy, Scar, and/or Sulcus Vocalis
Brief Title: Serial Platelet-Rich Plasma Injections for Vocal Fold Atrophy, Scar, and/or Sulcus Vocalis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Michael Johns, Professor, Otolaryngology-Head and Neck Surgery; Director, USC Voice Center, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APP-18-05224
Record Dates: First submitted 2018-09-29; First posted 2018-11-21 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-05

CONDITIONS: Presbylarynx; Atrophy; Larynx; Dysphonia; Vocal Cord Atrophy; Presbylarynges; Vocal Fold Scar; Sulcus Vocalis of Vocal Cord
Keywords: presbyphonia; presbylarynx; vocal fold atrophy; dysphonia; platelet rich plasma; PRP; vocal fold scar
MeSH Terms: conditions — Atrophy; Laryngeal Diseases; Dysphonia

STUDY DESIGN:
Intervention Model Description: Serial monthly vocal fold injections with PRP for total of 4 injections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serial PRP injections (Experimental): This arm will receive experimental intervention of serial monthly platelet-rich plasma (PRP) injections to a unilateral vocal fold mucosa for a total of 4 injections.
  Interventions: Procedure: Serial PRP injections

INTERVENTIONS:
Procedure: Serial PRP injections — Autologous platelet-rich plasma will be injected into the vocal fold mucosa in a serial fashion, once per month for a total of 4 injections.

SUMMARY:
This study will investigate the safety and efficacy of four serial monthly vocal fold injections of platelet-rich plasma to treat dysphonia secondary to vocal fold atrophy, scar, and/or sulcus vocalis with glottal insufficiency

DETAILED DESCRIPTION:
Vocal fold atrophy, scar, sulcus vocalis, glottal insufficiency with resulting dysphonia is a condition affecting millions of aging Americans, up to 35% of those 65 or older. Currently used treatment methods include voice therapy, injections of inert fillers, and laryngeal framework surgery. These modalities are imperfect with voice therapy requiring considerable time commitment, filler injections generally temporary in benefit, and surgery with increased risks. The investigators intend to conduct a single-arm study to assess the safety and efficacy of autologous platelet-rich plasma (PRP) injection for vocal fold atrophy, sulcus vocalis and scar. PRP is a substance purified from the patient's own blood that consists of platelets, growth factors, and other regenerative molecules that have been shown to promote rejuvenation in a variety of tissue types. Patients with vocal fold atrophy, sulcus vocalis, and scar identified in the USC Voice Center will be offered participation in a study to receive serial PRP injections in one vocal fold. Outcome measures evaluated pre- and post-injection and over follow-up visits will include various patient reported quality of life indices, objective clinical assessments of voice, and laryngeal videostroboscopy examinations. The investigators hypothesize that serial PRP injections will significantly improve vocal fold mucosal volume, morphology, and dysphonia in these patients with no adverse side effects.

ELIGIBILITY:
Inclusion Criteria:

* Vocal fold atrophy, scar, and/or sulcus vocalis diagnosed on laryngeal video stroboscopy by a fellowship-trained laryngologist
* Patients with a pre-injection VHI-10 score of ≥ 10
* Willingness to follow study requirements and perform follow-up visits for up to 4 months following the procedure
* Ability to give informed consent

Exclusion Criteria:

* Other co-existing laryngeal pathology that would affect either the safety or potential benefit from PRP injection
* Current smoker
* Underlying coagulopathy, thrombocytopenia, or platelet dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by FDA/CBER Adverse Event Severity Grading Scale | 4 months
  Adverse event severity grading scale from 1 to 4, with grade 1 as mild, grade 2 as moderate, grade 3 as severe, and grade 4 potentially life-threatening

SECONDARY OUTCOMES:
Voice-Related Quality of Life as assessed by Voice Handicap Index-10 (VHI-10) and Vocal Fatigue Index (VFI) | 4 months
  VHI-10 is a patient questionnaire with 10 statements rated from 0 to 4 with overall scale 0-40; VFI is a patient questionnaire with 19 statements rated from 0-4 with overall scale 0-76.
Objective Vocal Quality as assessed by experts using the Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) instrument | 4 months
  Blinded evaluations of audio voice recordings will be performed by laryngologists and speech-language pathologists using the CAPE-V, which grades overall severity, roughness, breathiness, strain, pitch, and loudness from 0-100.
Vocal Fold Appearance as assessed by experts using a modified version of the Voice-Vibratory Assessment with Laryngeal Imaging (VALI) form | 4 months
  Blinded assessments of recorded laryngeal videostroboscopy exams will be performed by laryngologists and speech-language pathologists using a modified version of the VALI, which is a graphical rating form to grade various components seen on stroboscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Johns, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradley JP, Hapner E, Johns MM 3rd. What is the optimal treatment for presbyphonia? Laryngoscope. 2014 Nov;124(11):2439-40. doi: 10.1002/lary.24642. Epub 2014 Aug 5. No abstract available. PMID 25132245
- [Background] Crawley BK, Dehom S, Thiel C, Yang J, Cragoe A, Mousselli I, Krishna P, Murry T. Assessment of Clinical and Social Characteristics That Distinguish Presbylaryngis From Pathologic Presbyphonia in Elderly Individuals. JAMA Otolaryngol Head Neck Surg. 2018 Jul 1;144(7):566-571. doi: 10.1001/jamaoto.2018.0409. PMID 29799925
- [Background] Cobden SB, Ozturk K, Duman S, Esen H, Aktan TM, Avunduk MC, Elsurer C. Treatment of Acute Vocal Fold Injury With Platelet-Rich Plasma. J Voice. 2016 Nov;30(6):731-735. doi: 10.1016/j.jvoice.2015.07.012. Epub 2015 Aug 17. PMID 26292799
- [Background] Woo SH, Jeong HS, Kim JP, Koh EH, Lee SU, Jin SM, Kim DH, Sohn JH, Lee SH. Favorable vocal fold wound healing induced by platelet-rich plasma injection. Clin Exp Otorhinolaryngol. 2014 Mar;7(1):47-52. doi: 10.3342/ceo.2014.7.1.47. Epub 2014 Feb 5. PMID 24587881
- [Background] Ozgursoy SK, Tunckasik F, Tunckasik ME, Akincioglu E, Dogan H, Beriat GK. Histopathologic Evaluation of Hyaluronic Acid and Plasma-Rich Platelet Injection into Rabbit Vocal Cords: An Experimental Study. Turk Arch Otorhinolaryngol. 2018 Mar;56(1):30-35. doi: 10.5152/tao.2018.2942. Epub 2018 Mar 1. PMID 29988271